CLINICAL TRIAL: NCT07397195
Title: Using Acceptance and Commitment Training to Promote Rehabilitation and Engagement in Values-Centered Living in Veterans Adapting to Inflammatory Bowel Disease and Mental Health Challenges (RECLAIM)
Brief Title: ACT for Veterans With IBD and Mental Health Challenges
Acronym: RECLAIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRD9-007-25M; 1IK2RD000689-01A2 (Other Grant/Funding Number: VA Office of Research and Development)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Inflammatory Bowel Diseases; Crohn's Disease; Ulcerative Colitis; Depressive Disorder; Anxiety Disorder; Stress Disorders, Post-Traumatic
Keywords: Acceptance and Commitment Therapy; Veterans; Inflammatory Bowel Diseases; Anxiety Disorders; Depressive Disorder; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Depressive Disorder; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RECLAIM (Experimental): One-day ACT group workshop tailored to the specific needs of Veterans with comorbid IBD and mental health conditions. This workshop focuses on teaching behavioral tools to help Veterans engage in values-driven behaviors when navigating difficult internal and external experiences.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Form of cognitive behavioral therapy that focuses on increasing psychological flexibility by fostering acceptance of difficult internal experiences, augmenting engagement in values-aligned behaviors, increasing contact with the present moment, and reducing reliance on avoidant coping.
  Other Names: ACT

SUMMARY:
Many Veterans with gastrointestinal disorders, such as inflammatory bowel disease (IBD), also have mental health conditions. IBD and mental health conditions can worsen one another through the brain-gut axis, leading to dramatic deficits in psychosocial functioning and quality of life (QOL). Yet, few Veterans with comorbid IBD and mental health conditions receive psychotherapy and no evidence-based psychotherapies have been tested in Veterans with these comorbidities. Adapting brief acceptance and commitment therapy (ACT) to the specific to the needs of these patients and embedding treatment into routine gastroenterology care may increase Veterans' access to efficient and effective rehabilitative care. This study aims to adapt and test an integrated, 1-Day ACT intervention tailored to the specific needs of Veterans with IBD and mental health conditions to improve psychosocial functioning and QOL.

DETAILED DESCRIPTION:
Nearly 80,000 Veterans have inflammatory bowel disease (Crohn's disease and ulcerative colitis; IBD). IBD is characterized by chronic inflammation of the gastrointestinal tract leading to significant pain, elimination difficulties, and functional impairment. Compounding these difficulties, nearly 50% of Veterans with IBD have comorbid depression, anxiety, and/or posttraumatic stress disorder. These comorbid conditions worsen IBD symptoms through the brain-gut axis, and lead to dramatic deficits in quality of life (QOL) and psychosocial functioning. Yet, less than 20% of patients with IBD and mental health conditions receive psychotherapy and 25-50% of psychotherapy patients drop out before clinically indicated. VA's integrated behavioral healthcare in primary and specialty care clinics increases therapy engagement and adherence, improving Veteran health and functioning. Despite this, psychogastroenterology services are underdeveloped in VA gastroenterology (GI) clinics. Moreover, no evidence-based psychotherapies have been tested in Veterans with comorbid IBD and mental health problems. It is essential to develop evidence-based psychotherapies for integrated use in GI clinics to practically increase access to care and improve the functioning and QOL of Veterans with GI conditions. Acceptance and commitment therapy (ACT) is a transdiagnostic psychotherapy that improves psychosocial functioning and QOL in patients with a variety of chronic and mental health conditions. ACT is flexibly delivered in various treatment formats, allowing providers to utilize methods that match the needs of specific populations and clinical settings. One-day ACT workshops improve access and retention while effectively and efficiently improving the psychosocial functioning of Veterans with various chronic health conditions. A pilot study of 1-day ACT for patients with IBD suggested preliminary feasibility, acceptability, and effectiveness in improving QOL. However, this pilot did not target Veterans or those with mental health conditions and was not delivered as an integrated part of GI care. This is a concern, as 1-day ACT is efficient and effective, yet is rarely used in routine clinical practice. Adapting 1-day ACT for integrated use in VA GI clinics will increase Veteran access to brief, evidence-based, rehabilitative treatment. This study aims to improve the psychosocial functioning and QOL of Veterans with comorbid IBD and mental health conditions by adapting and testing a 1-day, integrated ACT intervention, coined RECLAIM. The aims of this study are to: 1) Characterize the ACT-specific coping factors associated with psychosocial functioning and QOL in Veterans with IBD using survey and interview data to inform intervention adaptation; 2) Adapt a 1-day ACT intervention for Veterans with IBD and comorbid depressive, anxiety, and trauma disorders for integrated use in GI clinics. Pilot intervention (RECLAIM) with 10 Veterans and refine; 3) Test the feasibility and acceptability of RECLAIM with 40 Veterans with IBD and comorbid depressive, anxiety, and trauma disorders using a convergent mixed-methods design.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD as confirmed by the medical record
* Current diagnosis of a depressive, anxiety, or trauma-related disorder

Exclusion Criteria:

* Severe IBD symptoms that would prevent full participation in the study (i.e., hospitalized in the past 30 days, surgery in the past 30 days)
* Significant cognitive impairment
* Active suicidality
* Uncontrolled psychosis or bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2028-01-01 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | 2 week follow up
  Questionnaire evaluating patient perceptions of intervention feasibility
Therapist Fidelity to Treatment | Immediate post-therapy assessment
  Standardized rating tool assessing therapist fidelity to treatment protocol
Recruitment and Attrition Rates | Screening, baseline, Immediate post-therapy assessment, 2 week follow up, 3 month follow up, 6 month follow up
  Number of patients screened, approached, consented, completed treatment, and completed follow up assessment
Single item assessing participant engagement in treatment as rated by therapist | Immediate post-therapy assessment
  Assessment of participant treatment engagement
Percentage of treatment a patient completed | Immediate post-therapy assessment
  Assessment of participant treatment adherence
Acceptability of Intervention Measure (AIM) | 2 week follow up
  Questionnaire evaluating patient perceptions of the acceptability of treatment
Intervention Appropriateness Measure (IAM) | 2 week follow up
  Questionnaire evaluating patient perceptions of the appropriateness of treatment
Inflammatory Bowel Disease Questionnaire (IBDQ) | 3 month follow up
  Questionnaire evaluating IBD-specific quality of life
PROMIS-SF Social Functioning Scales | 3 month follow up
  Questionnaire evaluating participation in social roles, satisfaction with social roles, and social isolation
PROMIS-SF Psychosocial Illness Impact | 3 month follow up
  Questionnaire evaluating the psychosocial impact of chronic illness

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 (GAD-7) | 3 month follow up
  Questionnaire evaluating symptoms of anxiety
Patient Health Questionnaire- 9 (PHQ-9) | 3 month follow up
  Questionnaire evaluating depressive symptoms
PTSD Checklist for DSM-5 (PCL-5) | 3 month follow up
  Questionnaire evaluating symptoms of posttraumatic stress disorder
Visceral Sensitivity Index (VSI) | 3 month follow up
  Questionnaire evaluating GI-specific anxiety
Patient Reported Outcomes 2 and 3 (PRO2, PRO3) | 3 month follow up
  Questionnaire evaluating patient reported IBD symptoms
The Brief Pain Inventory-Short Form (BPI-SF) | 3 month follow up
  Questionnaire evaluating pain intensity and interference
Acceptance and Action Questionnaire-II (AAQ-II) | 3 month follow up
  Questionnaire evaluating psychological flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie Lynmarie Shanahan, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No